CLINICAL TRIAL: NCT06294834
Title: Improving Clinician Capacity to Provide Interventions for Manual Wheelchair Users
Acronym: SKILL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Dalhousie University (Other); National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lynn Worobey, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY22010071; 90SIMS0010 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2024-02-27; First posted 2024-03-06 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Paraplegia; Paralysis, Legs
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, two-period cross-over study design for Groups 1 and 2. Participants will complete baseline assessments and then be randomized to either Group 1 or Group 2. After enrollment for Groups 1 and 2 is complete, participants will be enrolled into Group 3.
Who Masked: Participant
Masking Description: For therapists, we will use a randomized, single-blinded, two-period cross-over study design for Groups 1 and 2. Participants will complete baseline assessments and then be randomized to either Group 1 or Group 2. After we have completed enrollment for Groups 1 and 2 we will enroll participants into Group 3.
  Rehabilitation professionals who are not therapists will be enrolled in Group 4.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: therapists (Other): Group 1 will receive the active intervention (intervention A) of remote wheelchair skills training. They will cross-over to receive the control intervention (intervention B) of education on wheelchair provision at 6 months.
  Interventions: Other: Part 1 of intervention A - Wheelchair skills training modules; Other: Part 2 of intervention A - Asynchronous feedback from a remote trainer; Other: Intervention B: Education on wheelchair provision
- Group 2 (Other): Group 2 will complete the control intervention (intervention B) of education on wheelchair provision. They will cross-over to receive the active intervention (intervention A) of remote wheelchair skills training at 6 months.
  Interventions: Other: Part 1 of intervention A - Wheelchair skills training modules; Other: Part 2 of intervention A - Asynchronous feedback from a remote trainer; Other: Intervention B: Education on wheelchair provision
- Group 3 (Other): Groups 3 will mirror Group 1 but for intervention A will only complete Part 1 of the training and then be cued weekly to practice.
  Interventions: Other: Part 1 of intervention A - Wheelchair skills training modules; Other: Intervention B: Education on wheelchair provision
- Group 4: rehab professionals, not therapists (Other): Group 4 will mirror Group 3 but receive access to both interventions at the same time.
  Interventions: Other: Part 1 of intervention A - Wheelchair skills training modules; Other: Intervention B: Education on wheelchair provision

INTERVENTIONS:
Other: Part 1 of intervention A - Wheelchair skills training modules — Clinicians will review a suite of training videos in a prescribed order that discuss motor learning principles, safe spotting, and how to complete 15 intermediate and advanced skills:
  1. Opening/closing doors
  2. getting over a gap
  3. getting over a threshold
  4. ascending a low curb
  5. descending a low curb
  6. ascending a high curb
  7. descending a high curb
  8. performing a stationary wheelie
  9. descending a high curb in a wheelie position
  10. descending a steep incline in a wheelie position and stopping
  11. ascending stairs
  12. descending stairs
  13. completing a floor-to-chair transfer
  14. car transfers
  15. folding and unfolding wheelchair
Other: Part 2 of intervention A - Asynchronous feedback from a remote trainer — Participants will practice of wheelchair skills paired with remote feedback. Participants will be reminded to practice once per week. The participant will practice any number of the 15 skills for a self-selected duration. Following each practice session, the participant will upload video(s) of the skills practiced and a session log, indicating any difficulties they encountered. The remote trainer will then review the video-recordings and reply to the participant with feedback.
  Arms: Group 1: therapists; Group 2
Other: Intervention B: Education on wheelchair provision — Participants will be provided with access to web-based wheelchair provision education modules. When the content is viewed will be self-selected by participants. Participants will be asked to complete a feedback survey at the end of the modules. Participants will receive weekly reminders to complete the intervention until a feedback survey completed.

SUMMARY:
The objective of this study is to determine the effectiveness of remote manual wheelchair skills training program for clinicians. The study will use three-group approach: intervention with remote feedback (Group 1), control group (Group 2), and structured self-study (Group 3). This demonstrates how the intervention compares not only to a control, but also to the next "best alternative" - therapists sourcing web-based training materials and learning independently.

DETAILED DESCRIPTION:
A randomized, single-blinded, two-period cross-over study design for Groups 1 and 2 will be used. Participants will complete baseline assessments and then be randomized to either Group 1 or Group 2. After enrollment for Groups 1 and 2 is completed, Group 3 participants will be enrolled.

Group 1 will receive the active intervention (intervention A) which will include a two-part training in wheelchair skills. For Part 1, they will review approximately 4 hours of educational videos on how to complete and teach wheelchair skills. For Part 2 they will complete a practice-feedback loop with a remote trainer providing asynchronous feedback. Group 3 will mirror Group 1 but complete only Part 1 of the training. Group 2 will receive the control intervention (intervention B) participants will review approximately 4 hours of educational videos. Participants will have 8 weeks to complete either training program. Both groups will then complete follow-up at 2 and 6 months. Following this, participants will cross over to receive the other intervention (Group 1 and 3 will receive intervention B, Group 2 will receive intervention A) and complete follow-up at 8 and 12 months.

Additionally, rehabilitation professionals who are not therapists will be able to access the training through a structured self-study (Group 4). This group will receive access to both trainings with follow-up at 2 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Practicing rehabilitation professional whose client population includes wheelchair users.
2. Willing and able to attempt practicing wheelchair skills
3. Access to a spotter(s)
4. Access to an Internet-ready device with video capabilities.
5. Speaks English

Exclusion Criteria:

1) Confident in teaching (Self-Efficacy on Assessing, Training, and Spotting [SEATS] item score = 5) and able to complete (WST-Q capacity item score = 2) >50% of skills targeted by the training intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Wheelchair Skills Test Questionnaire (WST-Q) score | baseline vs. 2 months
  Clinician capacity and confidence to complete wheelchair skills, as measured by wheelchair skills test questionnaire (WST-Q), will improve following training (Group 1,3) compared to the active control group (Group 2). The WST-Q includes values from 0-3 for each of Capacity, Confidence, and Performance. These three scores will be averaged. A higher value indicates a better outcome.
Change in Self-Efficacy on Assessing, Training, and Spotting (SEATS) score | baseline vs. 2 months
  Clinician confidence to provide wheelchair skills training, as measured by the Self-Efficacy on Assessing, Training, and Spotting (SEATS), will improve following training (Group 1,3) compared to the active control group (Group 2). The SEATS evaluation rates Assessing, Training, and Spotting, on scales from 0-5 for each skill. The values will be combined and averaged to assess progress over time. A higher score indicates improvement.
Change in number of wheelchair users trained | baseline vs. 6 months
  Clinician training of wheelchair users will increase in quantity (number of wheelchair users trained, duration of training) in the six months following training (Group 1,3) compared to the active control group (Group 2).
Change in quality of wheelchair skills trained | baseline vs. 6 months
  Clinician training of wheelchair users will increase in quality (number of wheelchair skills trained, capacity of trainees) in the year following training (Group 1,3) compared to the active control group (Group 2).

SECONDARY OUTCOMES:
Change in rehab professional Wheelchair Skills Test Questionnaire (WST-Q) score | baseline vs. 2 months, 6 months, and 1 year (Group 1,3 only) following training
  Rehabilitation professional capacity and confidence to complete wheelchair skills, as measured by wheelchair skills test questionnaire (WST-Q), will improve following training. The WST-Q includes values from 0-3 for each of Capacity, Confidence, and Performance. These three scores will be averaged. A higher value indicates a better outcome.
Change in rehab professional Self-Efficacy on Assessing, Training, and Spotting (SEATS) score | baseline vs. 2 months, 6 months, and 1 year (Group 1,3 only) following training
  Rehabilitation professional confidence to provide wheelchair skills training, as measured by the Self-Efficacy on Assessing, Training, and Spotting (SEATS), will improve following training. The SEATS evaluation rates Assessing, Training, and Spotting, on scales from 0-5 for each skill. The values will be combined and averaged to assess progress over time. A higher score indicates improvement.
Change in rehab professional quantity of wheelchair users trained | baseline vs. 6 months, and 1 year (Group 1,3 only) following training
  Rehabilitation professional training of wheelchair users will increase in quantity (number of wheelchair users trained, duration of training) following training.
Change in rehab professional quality of wheelchair training | baseline vs. 6 months, and 1 year (Group 1,3 only) following training
  Rehabilitation professional training of wheelchair users will increase in quality (number of wheelchair skills trained, capacity of trainees) in the year following training.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Worobey, PhD/DPT, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh / Rehab Neural Engineering Labs, Pittsburgh, Pennsylvania, United States